CLINICAL TRIAL: NCT06370715
Title: A 26- Week, Multicenter, Open-Label, Single-Arm, Phase 4 Study to Assess The Safety of Lyumjev in Adult Patients With Type 2 Diabetes Mellitus in India
Brief Title: A Study of LY900014 in Adult Participants With Type 2 Diabetes Mellitus in India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Cipla Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18269; I8B-MC-ITTA (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-04-15; First posted 2024-04-17 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes mellitus, type 2 diabetes, Lyumjev, basaglar, Humalog
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Insulin Lispro-aabc + Insulin Glargine (Experimental): Participants will receive insulin lispro-aabc in combination with insulin glargine administered by subcutaneous (SC) injection.
  Interventions: Drug: Insulin Lispro-aabc; Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Lispro-aabc — Administered SC
  Other Names: LY900014
Drug: Insulin Glargine — Administered SC

SUMMARY:
The purpose of this study is to assess the safety of insulin lispro-aabc in adult participants with Type 2 diabetes mellitus in India.

The study will last about 33 weeks for each participant, including screening (1 week), Lead-in period (4 weeks), treatment period (26 weeks) and follow up period (2 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 Diabetes Mellitus (T2DM) for ≥1 year prior to screening
* Treated for ≥90 days prior to screening with multiple daily injection (MDI) therapy

  * on basal insulin or insulin glargine 100 U/mL [Basaglar or Lantus] or insulin glargin 300 U/mL, insulin determir, insulin degludec U-100, or neutral protamine Hagedorn (NPH) insulin) in combination with at least 1 prandial injection of bolus insulin (insulin lispro 100 U/mL or 200 U/mL, insulin aspart, insulin glulisine, regular insulin, fast-acting insulin aspart), or
  * premixed analog or human insulin regimens with any basal and bolus insulin
* May have been treated with up to 3 oral antihyperglycemic medications (OAMs) including metformin, sodium-glucose cotransporter (SGLT)-2 inhibitor in accordance with local regulations. The dose of all OAMs must have been stable for ≥90 days prior to screening
* Have an HbA1c value ≥7.5% and ≤10% according to the central laboratory at screening
* Body mass index ≤45.0 kg/m²
* Have access to a telephone, or alternative means for close monitoring/communications
* Have refrigeration at home or have ready access to refrigeration for storage of insulin therapy
* Have a regular wake-sleep schedule (awake-work during the day and sleep during the night)

Exclusion Criteria:

* Having any other condition (including known drug or alcohol abuse, psychiatric disorder including eating disorder) that precludes the subject from following and completing the protocol
* Have been diagnosed, at any time, with type 1 diabetes mellitus (T1DM) or latent autoimmune diabetes in adults
* Have hypoglycemia unawareness as judged by the investigator
* Have had any episode of severe hypoglycemia (defined as requiring assistance due to neurologically disabling hypoglycemia) within the 6 months prior to screening
* Have had 1 or more episodes of diabetic ketoacidosis or hyperglycemic hyperosmolar state within the 6 months prior to screening
* Have a known diagnosis of secondary diabetes (for example, diabetes caused by hemochromatosis, acromegaly, chronic pancreatitis, or pancreatectomy)
* Excessive insulin resistance defined as having received a total daily dose of insulin >2.0 U/kg at the time of screening
* Have a history of or are being evaluated for bariatric surgery including Roux-en-Y gastric bypass surgery, gastric banding, and/or gastric sleeve
* Have cardiovascular disease, within the past 6 months prior to screening, defined as stroke, decompensated heart failure (New York Heart Association Class III or IV), myocardial infarction, unstable angina pectoris, or coronary arterial bypass graft
* History of renal transplantation
* Currently receiving renal dialysis
* Serum creatinine >2.0 mg/dL (177 µmol/L) at screening
* Have obvious clinical signs or symptoms of liver disease (for example, acute or chronic hepatitis or cirrhosis), or elevated liver enzyme measurements
* Have active or untreated malignancy, have been in remission from clinically significant malignancy (other than basal cell or squamous cell skin cancer) for less than 5 years, or are at an increased risk for developing cancer or a recurrence of cancer in the opinion of the investigator
* Have had a blood transfusion or severe blood loss within 90 days prior to screening or have known hemoglobinopathy, anemia, or any other traits known to interfere with measurement of HbA1
* Have presence of clinically significant gastrointestinal disease (for example, clinically active gastroparesis associated with wide glucose fluctuations) in the investigator's opinion
* Have used thiazolidinediones, glucagon-like peptide 1 receptor agonist, or pramlintide within 90 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with at least 1 Episode of Hypoglycemia | Baseline through Week 26
  Percentage of participants with at least 1 episode of hypoglycemia will be reported.

SECONDARY OUTCOMES:
Percentage of Participants with Severe Hypoglycemic Events | Week 26
  Percentage of participants with severe hypoglycemic events defined as (events/participants/year).
Percentage of Participants with Nocturnal Hypoglycemia Events | Week 26
  Percentage of participants with nocturnal hypoglycemia events defined as the incidence and rate (events/participant/year) of nocturnal hypoglycemia (BG<54 mg/dL).
Percentage of Participants with Nocturnal and All Documented Hypoglycemic Events | Week 26
  Percentage of participants with nocturnal and documented hypoglycemia events will be reported.
Change from Baseline to Week 26 in Body Weight | Baseline, Week 26
  Change from baseline to week 26 in body weight will be reported.
Change from Baseline to Week 26 in Insulin Treatment Satisfaction Questionnaire (ITSQ) Score | Baseline, Week 26
  The ITSQ is a 22-item, participant-completed questionnaire that assesses insulin treatment satisfaction over the past 4 weeks for participants with diabetes in 5 domains: Inconvenience of Regimen (5 items), Lifestyle Flexibility (3 items), Glycemic Control (3 items), Hypoglycemic Control (5 items), Insulin Delivery Device Satisfaction (6 items). Participants respond to each item on a 7-point Likert scale ranging from "not at all" to "extremely." Scores can be generated for each domain and the overall score is transformed to a scale of 0-100. Higher scores indicate better treatment satisfaction.
Change from Baseline to Week 26 in Hemoglobin A1c (HbA1c) | Baseline, Week 26
  Change from baseline to week 26 in HbA1c will be reported.
Percentage of Participants Achieving HbA1c Less Than (<) 7% | Week 26
  Percentage of participants achieving HbA1c <7% will be reported.
Change from Baseline to Week 26 in 1- and 2-hour Postprandial Glucose (PPG) Values | Baseline, Week 26
  1- and 2-hour PPG values are estimated from self-monitored blood glucose (SMBG)
Change from Baseline to Week 26 in Bolus Insulin Dose | Baseline, Week 26
  Change from Baseline to Week 26 in Bolus Insulin Dose will be reported.
Change from Baseline to Week 26 in Basal Insulin Dose | Baseline, Week 26
  Change from Baseline to Week 26 in Basal Insulin Dose will be reported.
Change from Baseline to Week 26 in Bolus Basal: Bolus Ratio | Baseline, Week 26
  Change from Baseline to Week 26 in Basal: Bolus Ratio will be reported.
Change from Baseline to Week 26 in 9-Point Self-Monitored Blood Glucose (SMBG) Values | Baseline, Week 26
  SMBG measurements were taken at 9 time points: fasting, 1 hour post breakfast, 2 hours post breakfast, pre lunch,1 hour post lunch, 2 hours post lunch, pre dinner, 1 hour post dinner, and 2 hours post dinner.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- India (12):
  - Osmania Medical College & Hospital, Hyderabad, Andhra Pradesh
  - King George Hospital, Visakhapatnam, Visakhapatnam, Andhra Pradesh
  - Diabetes Research Centre, Royapuram, Chennai India
  - Vijyaratna Dibetes Diagnosis Treatment Centre, Ahmedabad, Gujarat
  - Center for Diabetes and Endocrine Care, Bengaluru, Karnataka
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Chellaram Diabetes Institute, Pune, Maharashtra
  - S. P. Medical College & A G Hospital, Bikaner, Rajasthan
  - Rajasthan University of Health Sciences, Jaipur, Rajasthan
  - Kovai Diabetes Speciality Center and Hospital, Coimbatore, Tamil Nadu
  - Brij Medical Center Pvt. Ltd., Kanpur, Uttar Pradesh
  - Medical College & Hospital, Kolkata, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/